CLINICAL TRIAL: NCT03767920
Title: Role of Co-administered Dexamethasone in Transversus Abdominis Plane Block After Cesarean Section: A Randomized, Double-blind Controlled Trial
Brief Title: Role of Dexamethasone in Transversus Abdominis Plane Block After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/180/7/18
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section
Keywords: dexamethasone; transversus abdominis plane block; cesarean section
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A prospective Randomized Interventional double-blind study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participating patients, surgeons, anesthesiologists and medical investigators who will be involved in the data collection will be all blinded to the patient's group assignment until the collection of data for all cases will be complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine and dexamethasone (Active Comparator): Bilateral TAP block with 20 ml of 0.25% bupivacaine + 4 mg/kg dexamethasone diluted with isotonic saline.
  Interventions: Drug: bupivacaine; Drug: dexamethasone
- bupivacaine and placebo to dexamethasone (Active Comparator): BilateralTAP block with 20 ml of 0.25% bupivacaine bilaterally plus placebo to dexamethasone
  Interventions: Drug: bupivacaine; Drug: placebo to dexamethasone

INTERVENTIONS:
Drug: bupivacaine — TAP block with 20 ml of 0.25% bupivacaine bilaterally
  Other Names: Active Comparator
Drug: dexamethasone — TAP block with 4 mg dexamethasone bilaterally
  Other Names: active comparator
  Arms: bupivacaine and dexamethasone
Drug: placebo to dexamethasone — TAP block with 4 mg placebo to dexamethasone bilaterally
  Other Names: Placebo
  Arms: bupivacaine and placebo to dexamethasone

SUMMARY:
Our aim to study the efficacy of bupivacaine 0.25% with dexamethasone and that of bupivacaine 0.25% alone in transversus abdominis plane (TAP) block for postoperative analgesia in patients undergoing an elective Caesarean section.

* Group 1: bupivacaine 0.25% + dexamethasone 8 mg
* Group 2: bupivacaine 0.25% A prospective Randomized Interventional double-blind study.

DETAILED DESCRIPTION:
The pain and discomfort following cesarean delivery are mostly due to the abdominal wall incision and dissection of muscles; it delays early ambulation and breastfeeding. This can lead to postoperative complications such as thromboembolic disorders. So, providing an effective and safe postoperative analgesic method seems to be mandatory. Opioid analgesia remains the most effective means of relieving pain in a wide variety of conditions; however, it may cause adverse effects such as nausea, vomiting, pruritus, urinary retention, and respiratory depression. As the analgesia and the side effects of opioids are dose-dependent, a multimodal approach may enhance analgesia, which in turn would decrease the side effects .

Mc Donnell and colleagues have reported that a transversus abdominis plane (TAP) block can decrease the postoperative pain following abdominal surgery. The landmarks of this block were first described in 2001 by Rafi. The TAP block has been performed for postoperative analgesic control in patients undergoing radical prostatectomy, hysterectomy, cesarean delivery under spinal anesthesia, and laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* healthy parturient (ASA I and II) scheduled to undergo LSCS under spinal anesthesia

Exclusion Criteria:

* Participants had known sensitivity to bupivacaine
* patient refusal,
* localized infection over injection point
* patients with significant coagulopathies and
* with contraindications to regional anesthesia,
* patients with heart diseases, altered renal or liver functions,
* psychological disorders, patients with pregnancy-induced hypertension and
* gestational diabetes, chronic use of pain medications,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — healthy parturient scheduled to undergo LSCS under spinal anesthesia
Enrollment: 120 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score for pain during movement | 6 hours post operative
  movement-evoked pain measurements ranging from 0 to 10, where 0 no pain and 10 maximum pain

SECONDARY OUTCOMES:
Visual analog score during rest | 48 hours postoperative
  ranging from 0 to 10, where 0 no pain and 10 maximum pain
number of patients need Fentanyl consumption | 48 hours postoperative
  number of patients need Fentanyl consumption
number of days patients stay in hospital | 4 weeks
  calculation of number of days patients stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No